CLINICAL TRIAL: NCT00211432
Title: Treatment of Pseudovitellium Detachment With Open-Label Anecortave Acetate Sterile Suspension (15 mg)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Joan, Lawrence A. Yannuzzi, M.D., Manhattan Eye, Ear & Throat Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pseudovitellium Detachment
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Pseudovitellium Detachment; Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Title: Treatment of Pseudovitellium Detachment (Experimental): Open-Label Anecortave Acetate Sterile Suspension(15mg)
  Interventions: Drug: Anecortave Acetate Sterile Suspension (15 mg)

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension (15 mg)

SUMMARY:
The purpose of this study is to provide compassionate use of anecortave acetate sterile suspension of 15 mg for a series of five patients as a means to control pseudovitelliform detachment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of patients with pseudovitellium detachment.
2. Patients must be at least 18 years of age.
3. Visual acuity of 20/30 to 20/320 in study eye on the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity chart
4. Visual acuity of 20/800 or better in fellow eye on the ETDRS visual acuity chart

Exclusion Criteria:

1. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
2. Patients who have undergone intraocular surgery within the last 2 months.
3. Patient participating in any other investigational drug study.
4. Use of an investigational drug or treatment related or unrelated to their condition within 30 days prior to receipt of study medication.
5. Inability to obtain photographs to document choroidal neovascularization (CNV) (including difficulty with venous access).
6. Patient with significant liver disease or uremia.
7. Patient with known adverse reaction to fluorescein and indocyanine green or iodine.
8. Patient has a history of any medical condition which would preclude scheduled visits or completion of study
9. Patient has had insertion of scleral buckle in the study eye
10. Patient has received radiation treatment
11. Patient is on anticoagulant therapy with the exception of aspirin
12. Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Title: Treatment of Pseudovitellium Detachment With Open-Label Anecortave Acetate Sterile Suspension (15mg) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Yannuzzi, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States